CLINICAL TRIAL: NCT01797029
Title: A Randomized, Double-Blind, Placebo-Controlled Trial on the Clinical Efficacy and Safety of a Single Dose of Trivalent Seasonal Live-Attenuated Influenza Vaccine(LAIV) Among Children Aged 24 Through 59 Months in Bangladesh
Brief Title: A Randomized, Controlled Trial on the Efficacy and Safety of Live-Attenuated Influenza Vaccine (LAIV) Among Children in Bangladesh
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PATH (Other)
Collaborators: Johns Hopkins University (Other); International Centre for Diarrhoeal Disease Research, Bangladesh (Other); Centers for Disease Control and Prevention (U.S. Federal Agency); Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LAIV-CE-01
Record Dates: First submitted 2013-02-20; First posted 2013-02-22 (Estimated); Results first posted 2015-05-15 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2014-07

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vaccine (Experimental)
  Interventions: Biological: SIIL Live Attenuated Influenza Vaccine
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: SIIL Live Attenuated Influenza Vaccine — A single dose of SIIL Trivalent LAIV--2012/2013 Northern Hemisphere vaccine containing A/California/7/2009 (H1N1), A/Victoria/361/2011 (H3N2), B/Wisconsin/1/2010
  Arms: Vaccine
Biological: Placebo — A single dose of inactive placebo will be identical to reconstituted SIIL LAIV in ingredients and concentrations except A/California/7/2009 (H1N1), A/Victoria/361/2011 (H3N2), B/Wisconsin/1/2010 will be replaced with egg allantoic fluid.
  Arms: Placebo

SUMMARY:
This is a single center, multi-site, double-blind, parallel group, placebo-controlled trial of the clinical efficacy of trivalent Serum Institute of India, Ltd. (SIIL)live-attenuated influenza vaccine (LAIV) vaccine among children aged 24 through 59 months in Bangladesh.

Background:

1. Burden: Within Bangladesh, community- based influenza surveillance identified 84.5 cases/1000 children-years among children <5 years, while 10% of clinical pneumonia cases were influenza positive in this age group.
2. Knowledge gap: There has never been a randomized clinical efficacy trial of the SIIL LAIV vaccine conducted among children in a low-income country.
3. Relevance: Another LAIV vaccine (made by MedImmune) has been shown to have high efficacy against laboratory-confirmed influenza among children. The SIIL LAIV has the potential to be an inexpensive intervention to prevent pediatric influenza disease.

Primary Hypothesis: In children aged 24 through 59 months in Bangladesh, LAIV is efficacious in reducing rates of symptomatic, laboratory-confirmed influenza (vaccine-matched strains) among children vaccinated with LAIV as compared to children vaccinated with a placebo through the first influenza season following vaccination.

Primary Objective: To determine the efficacy of LAIV in reducing rates of symptomatic, laboratory-confirmed influenza virus infection (vaccine-matched strains) among children receiving LAIV as compared to children receiving a placebo through the first influenza season following vaccination (through December 2013).

Methods: A total of 1761 children will be enrolled and randomized in a 2:1 ratio of LAIV to placebo beginning in March 2013. After vaccination, all children will be evaluated for reactions with one home visit four days post vaccination. Subsequently, all children will be monitored weekly for safety outcomes and illness signs at weekly field worker home visits through December 2013. An extended surveillance period was added to this study and, for participants consenting to additional follow-up, surveillance will extend through a second season (through September 2014). Participants with illness signs will be referred to the study clinic for evaluation using standardized diagnostic criteria and treatment by a study physician. Children meeting protocol-defined clinical Specimen Collection Criteria will have a nasopharyngeal wash specimen collected. Clinical specimens will be tested by Real time polymerase chain reaction (rRT-PCR) for evidence of influenza virus infection.

Primary Outcome measures/variables: Vaccine efficacy will be assessed against symptomatic, laboratory-confirmed influenza for all circulating virus strains.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female child at least 24 months of age and no older than 59 months of age at the time of study vaccination.
* A child whose parent or guardian's primary residence, at the time of study vaccinations, is within the Kamalapur surveillance site catchment area or Matlab service area and who intends to be present in the area for the duration of the trial.
* A child whose parent or legal guardian is willing to provide written informed consent prior to the participant's study vaccination.

Exclusion Criteria:

* Has any serious, active, medical conditions, including: a chronic disease of any body system, chronic infections such as tuberculosis, genetic disorders, such as Down's syndrome or other cytogenetic disorder, known or suspected disease of the immune system.
* Is receiving immunosuppressive agents, including systemic corticosteroids, during the month prior to study vaccination.
* Has a history of documented hypersensitivity to eggs or other components of the vaccine (including gelatin, sorbitol, lactalbumin and chicken protein), or with life-threatening reactions to previous influenza vaccinations.
* Has ever received influenza vaccine (LAIV or inactivated).
* History of Guillain-Barre syndrome
* Is receiving aspirin therapy or aspirin-containing therapy currently or two weeks before.
* Lives in household with somebody currently participating in a respiratory vaccination or antiviral study.
* Has current or past participation (within 2 months of trial enrollment visit) in any clinical trial involving a drug or biologic with activity against respiratory disease.
* History of a previous severe allergic reaction with generalized urticarial, angioedema, or anaphylaxis.
* Has any condition determined by investigator as likely to interfere with evaluation of the vaccine or be a significant potential health risk to the child or make it unlikely that the child would complete the study

Temporary Inclusion Contraindications:

* Concurrent febrile illness (measured temperature 38 degrees C axillary).
* Active wheezing illness

Ages: 24 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1761 (Actual)
Dates: Start 2013-02; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abdullah Brooks, MD, MPH, Principal Investigator — Johns Hopkins University
Locations (2):
- Bangladesh (2):
  - icddr, b Kamalapur, Dhaka
  - icddr,b Matlab, Matlab

REFERENCES:
- [Derived] Rotrosen E, Zaman K, Feser J, Ortiz JR, Goswami D, Sharmeen AT, Rahman M, Lewis KDC, Rahman MZ, Barin B, Brooks WA, Neuzil KM. Influenza Among Young Children in Bangladesh: Clinical Characteristics and Outcomes From a Randomized Clinical Trial. Clin Infect Dis. 2017 Nov 13;65(11):1914-1920. doi: 10.1093/cid/cix674. PMID 29028980
- [Derived] Brooks WA, Zaman K, Lewis KD, Ortiz JR, Goswami D, Feser J, Sharmeen AT, Nahar K, Rahman M, Rahman MZ, Barin B, Yunus M, Fry AM, Bresee J, Azim T, Neuzil KM. Efficacy of a Russian-backbone live attenuated influenza vaccine among young children in Bangladesh: a randomised, double-blind, placebo-controlled trial. Lancet Glob Health. 2016 Dec;4(12):e946-e954. doi: 10.1016/S2214-109X(16)30200-5. Epub 2016 Oct 13. PMID 27746226

RESULTS

PARTICIPANT FLOW:
Groups:
- Vaccine: A single dose of Serum Institute of India, Ltd. (SIIL) Trivalent LAIV--2012/2013 WHO Northern Hemisphere vaccine containing A/California/7/2009 (H1N1), A/Victoria/361/2011 (H3N2), B/Wisconsin/1/2010
- Placebo: Inactive placebo will be identical to reconstituted Serum Institute of India, Ltd. (SIIL) LAIV in ingredients and concentrations except A/California/7/2009 (H1N1), A/Victoria/361/2011 (H3N2), B/Wisconsin/1/2010 will be replaced with egg allantoic fluid.
Period: Overall Study
Arm/Group | Vaccine | Placebo
Started | 1174 | 587
Completed | 1015 | 526
Not Completed | 159 | 61

BASELINE CHARACTERISTICS:
Population: All participants receiving the single dose of study vaccination.
Groups:
- Vaccine: A single dose of SIIL Trivalent LAIV--2012/2013 WHO Northern Hemisphere vaccine containing A/California/7/2009 (H1N1), A/Victoria/361/2011 (H3N2), B/Wisconsin/1/2010
- Placebo: Inactive placebo will be identical to reconstituted SIIL LAIV in ingredients and concentrations except A/California/7/2009 (H1N1), A/Victoria/361/2011 (H3N2), B/Wisconsin/1/2010 will be replaced with egg allantoic fluid.
- Total: Total of all reporting groups
Arm/Group | Vaccine | Placebo | Total
Number analyzed (Participants) | 1174 | 587 | 1761
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1174 | 587 | 1761
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 589 | 306 | 895
  Male | 585 | 281 | 866
Region of Enrollment [Number; unit: participants]
  Bangladesh | 1174 | 587 | 1761

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Symptomatic, Laboratory-confirmed Influenza Virus Infection (Vaccine-matched Strains).
Time Frame: Through 7 to 9 months post-vaccination
Measure: Number; unit: percentage of participants
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 1174 | 587
percentage of participants | 6.7 | 15.8
Statistical Analysis 1: Comparison: Vaccine vs Placebo; Test type: Superiority or Other; p < 0.0001, Fisher Exact

2. Secondary Outcome: Safety Profile of LAIV: Solicited and Unsolicited Local and Systemic Reactions
Time Frame: Through one week post-vaccination
Reporting Status: Not Posted

3. Secondary Outcome: Safety Profile of LAIV: Immediate Reactions
Time Frame: 30 minutes post-vaccination
Measure: Number; unit: participants
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 1174 | 587
participants | 0 | 0

4. Secondary Outcome: Safety Profile of LAIV: Serious Adverse Events
Time Frame: Through 7 to 9 months post-vaccination
Reporting Status: Not Posted

5. Secondary Outcome: Safety Profile of LAIV: Protocol Defined Wheezing Illness
Time Frame: Through 7 to 9 months post-vaccination
Reporting Status: Not Posted

6. Secondary Outcome: Percentage of Participants With Symptomatic, Laboratory-confirmed, Influenza Virus Infection (All Strains)
Time Frame: Through 7 to 9 months post-vaccination
Reporting Status: Not Posted

7. Secondary Outcome: The Clinical Characteristics of Influenza, Including Influenza Co-infections With Other Bacterial and Viral Respiratory Pathogens
Time Frame: Through 16 to 19 months post-vaccination
Reporting Status: Not Posted

8. Secondary Outcome: The Viral Etiologies of Acute Respiratory and Febrile Illness
Time Frame: Through 16 to 19 months post-vaccination
Reporting Status: Not Posted

9. Secondary Outcome: Safety Profile of LAIV: Serious Adverse Events
Time Frame: Through 16 to 19 months post-vaccination
Reporting Status: Not Posted

10. Secondary Outcome: Safety Profile of LAIV: Protocol Defined Wheezing Illness
Time Frame: Through 16 to 19 months post-vaccination
Reporting Status: Not Posted

11. Secondary Outcome: Percentage of Participants With Symptomatic, Laboratory-confirmed, Influenza Virus Infection (All Strains)
Time Frame: Through 16 to 19 months post-vaccination
Reporting Status: Not Posted

12. Secondary Outcome: Percentage of Participants With Symptomatic, Laboratory-confirmed Influenza Virus Infection (Vaccine-matched Strains).
Time Frame: Through 16 to 19 months post-vaccination
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Percentage of Participants With Moderate to Severe, Laboratory-confirmed Influenza Virus Infection Among Children
Time Frame: Through 7 to 9 months post-vaccination
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Percentage of Participants With Moderate to Severe, Laboratory-confirmed Influenza Virus Infection Among Children
Time Frame: Through 16 to 19 months post-vaccination
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Percentage of Participants With Symptomatic, Laboratory-confirmed Influenza Virus Infection (Vaccine-matched Strains) Among Children
Time Frame: From approx. 6 months to approximately 19 months post-vaccination
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Percentage of Participants With Symptomatic, Laboratory-confirmed Influenza Virus Infection (All Strains) Among Children
Time Frame: From approx. 6 months to approximately 19 months post-vaccination
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Throughout study period: February 2013 to September 2014, up to 20 months of follow-up.
Description: Adverse events are classified according to the type of adverse event.
Arm/Group | Vaccine | Placebo
Serious Adverse Events (participants affected / at risk) | 42/1174 | 19/587
Other Adverse Events (participants affected / at risk) | 68/1174 | 35/587
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vaccine (N=1174) | Placebo (N=587)
Respiratory SAEs (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 8 (8)
Non respiratory SAEs (General disorders) | 31 (31) | 11 (11)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vaccine (N=1174) | Placebo (N=587)
Any SOC (General disorders) | 68 | 35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less